CLINICAL TRIAL: NCT06282796
Title: Early Prediction and Warning for Cardiotoxicity Due to Anthracycline-Based Breast Cancer Chemotherapy: a Prospective, Multicenter, Clinical Trial
Brief Title: Early Prediction and Warning for Cardiotoxicity Due to Anthracycline-Based Breast Cancer Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: EPW-CABC-01
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Chemotherapy; Anthracyclines; Cardiotoxicity; Early detection
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anthracycline-Based Breast Cancer Chemotherapy Group: Age ≥18 years, histologically or cytopathologically confirmed stage I-III HER2+ breast cancer, scheduled to receive consecutive anthracycline chemotherapy or subsequent sequential trastuzumab targeted therapy, with a prechemotherapy LVEF≥53%.
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — Two-dimensional, color Doppler, spectral Doppler, tissue Doppler and three-dimensional echocardiographic image recordings will be taken using a Philips Epiq 7C echocardiography device and X5-1 probe. Conventional parameters, additional parameters, and strain analyzes will be performed by TomTec AutoStrain Suite Software

SUMMARY:
This multicenter clinical study aims to build an intelligent and accurate diagnosis and dynamic prediction and early warning model of cardiotoxicity due to anthracycline-based breast cancer chemotherapy, clarify the value of the early warning model in guiding the targeted prevention of myocardial protection, providing an important theoretical basis for reducing the mortality rate of breast cancer and improving the prognosis.

DETAILED DESCRIPTION:
The latest global cancer burden data released by the World Health Organization International Agency for Research on Cancer (IARC) has shown that the incidence of breast cancer ranks first in the world. Anthracycline-based treatments are first-line chemotherapy agents to treat early breast cancer. Although anthracycline-based treatments has significantly improved the 5-year survival rate of breast cancer patients, the cancer therapy-related cardiac dysfunction (CTRCD) caused by anthracyclines has become the major cause of breast cancer death. However, CTRCD patients often have no obvious symptoms of heart failure in the early stage, and the diagnosis is very secretive, resulting in delayed intervention, unable to timely terminate the disease process, and seriously affecting the prognosis.

Echocardiography has the advantages of real-time, non-invasive and repeatable, and is the preferred detection method for asymptomatic CTRCD at present. The diagnosis of asymptomatic CTRCD depends on the change of left ventricular (LV) ejection fraction (EF) and global longitudinal strain (GLS) before and after chemotherapy. However, the measurement of LVEF and GLS is based on manual methods, resulting in poor repeatability. Cardiotoxicity due to anthracycline-based breast cancer chemotherapy progresses gradually and changes dynamically with dose and time.

Therefore, this study intends to build an intelligent model for early prediction and warning of asymptomatic CTRCD, so as to provide a reliable basis for timely adjustment of individualized cardiac protection strategies and maintaining LV function and reducing mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically or cytopathological confirmed stage I-III HER2+ breast cancer, scheduled to receive consecutive anthracycline chemotherapy or subsequent sequential trastuzumab targeted therapy
* LVEF≥53% before chemotherapy

Exclusion Criteria:

* life expectancy ≤12 months
* Participating in other ongoing oncology clinical trials
* Prior treatment with anthracyclines or chest radiation therapy
* Pregnant or lactating women
* Ultrasound images of the heart are of very poor quality

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with anthracycline-based breast cancer chemotherap
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction(unit: %) in all breast cancer patients treated with anthracycline-based chemotherapy. | 1 day after admission
  To Evaluate the changes of cardiac systolic function in all breast cancer patients treated with anthracycline-based chemotherapy.

SECONDARY OUTCOMES:
Left ventricular global longitudinal strain (unit: %) in all breast cancer patients treated with anthracycline-based chemotherapy. | 1 day after admission
  To Evaluate of the subclinical changes of cardiac systolic function in all breast cancer patients treated with anthracycline-based chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghuai Wang, Ph.D, Principal Investigator — the First Hospital of China Medical Univeristy
Locations (5):
- China (5):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Dalian Friendship Hospital, Dalian, Liaoning
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The Third People's Hospital Of Chengdu, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided